CLINICAL TRIAL: NCT07099378
Title: Relationship Between Micro Ribonucleic Acid (miRNA) Expression and Inflammatory Factors in Patients With Parkinson's and Periodontal Disease
Brief Title: Micro Ribonucleic Acid (miRNA) Expression and Inflammatory Factors in Patients With Parkinson's and Periodontal Disease
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, Melis Yilmaz, Assistant Prof Dr, Medipol University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 106
Record Dates: First submitted 2025-07-25; First posted 2025-08-01 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Periodontal Diseases Inflammation
Keywords: periodontal disease miRNA

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Comparator (Active Comparator): Collection of patients' saliva and serum and analysis of sample molecules.
  Interventions: Other: Saliva and Serum
- Experimental (Experimental): ELISA method will be used to measure TNF-α values in collected saliva and serum samples.RT-qPCR based miRNA gene expression analyses will be performed with 2-step qRT-PCR Kits (Thermofisher Scientific, MA, USA).
  Interventions: Other: Saliva and Serum

INTERVENTIONS:
Other: Saliva and Serum — Saliva were collected to analyze the selected markers as unstimulated samples during the early hours of the day. The saliva was centrifuged and then transferred into Eppendorf tubes. Venous puncture was performed after saliva collection and 10 mL of blood samples were collected by qualified staff from each participant.Saliva and serum were then stored at -80 °C until analysis.
  Arms: Active Comparator
Other: Saliva and Serum — ELISA method will be used to measure TNF-α values in collected saliva and serum samples.RT-qPCR based miRNA gene expression analyses will be performed with 2-step qRT-PCR Kits (Thermofisher Scientific, MA, USA).
  Arms: Experimental

SUMMARY:
MicroRNAs are important regulators of the immune and inflammatory response to bacterial pathogens during periodontal disease.The aim of this study was to evaluate the possible miRNA type for Parkinson's in saliva of orally healthy individuals.

DETAILED DESCRIPTION:
A total of 51 individuals, 35 systemically healthy and 16 with Parkinson's disease and both dental and periodontal health, were included in the study.Clinical periodontal parameters, DMFT data and salivary flow rates were recorded.Unstimulated saliva samples were taken from each participant and miRNA was evaluated by RT-qPCR method.ELISA method was used to measure TNF α values in collected saliva and serum samples.

ELIGIBILITY:
Inclusion Criteria:

* dentally and periodontally healthy

  * Systemically healthy with no uncontrolled chronic and/or autoimmune disease
  * No systemic, neurological, or autoimmune disease in addition to Parkinson's disease.

Exclusion Criteria:

* history of regular use of systemic antibiotics anti-inflammatory, or antioxidant drugs (previous 3 months)
* nonsurgical periodontal treatment (previous 6 months)
* surgical periodontal treatment (previous 12 months)
* presence of<20 teeth
* current medications affecting gingival health (calcium channel blockers, phenytoin, cyclosporine, and hormone replacement therapy)
* diabetes
* diagnosis of rheumatoid arthritis
* pregnancy
* lactating
* smoking
* excessive alcohol consumption.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 51 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
1. Pocket probing depth | 6 months
  Measurement of the depth of a sulcus or periodontal pocket determined by measuring distance from a gingival margin to the base of the sulcus or pocket with a calibrated periodontal probe.
2.Clinical attachment level | 6 months
  Clinical attachment level (or loss, CAL) is a more accurate indicator of the periodontal support around a tooth than probing depth alone. CAL is measured from a fixed point on the tooth that does not change, the CEJ.
  To calculate CAL, two measurements are needed: distance from the gingival margin to the CEJ and probing depth.
  In recession: probing depth (+) gingival margin to the CEJ (add). In tissue overgrowth: probing depth (-) gingival margin to the CEJ (subtract)
3.Bleeding on probing | 6 months
  referring to bleeding that is induced by gentle manipulation of the tissue at the depth of the gingival sulcus, or interface between the gingiva and a tooth.

SECONDARY OUTCOMES:
4.Saliva and serum samples processing and analyses | 1 month
  ELISA method will be used to measure TNF-α values in collected saliva and serum samples.RT-qPCR based miRNA gene expression analyses will be performed with 2-step qRT-PCR Kits (Thermofisher Scientific, MA, USA).

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Medipol University, Istanbul, Fatih, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No